CLINICAL TRIAL: NCT04894188
Title: Neoadjuvant Hormone and Radiation Therapy Followed by Radical Prostatectomy in Patients With High-Risk Locally Advanced Prostate Cancer and Biomarker Research
Brief Title: Neoadjuvant Hormone and Radiation Therapy Followed by Radical Prostatectomy in Patients With High-Risk Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202101088RINA
Record Dates: First submitted 2021-05-09; First posted 2021-05-20 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2021-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Goserelin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant RT and ADT (Experimental): Intensity modulated radiation therapy (IMRT), with 50 Gy in 25 daily fractions (2 Gy/fraction, 5 fractions weekly) for 5 weeks (week 1 - week 5).
  Gosereline 3.6mg sc injection at week 1, week 5, and week 9
  Interventions: Radiation: radiation therapy; Drug: Goserelin 3.6 MG; Procedure: radical prostatectomy
- Neoadjuvant ADT (Active Comparator): Gosereline 3.6mg sc injection at week 1, week 5, and week 9
  Interventions: Drug: Goserelin 3.6 MG; Procedure: radical prostatectomy

INTERVENTIONS:
Radiation: radiation therapy — Intensity modulated radiation therapy (IMRT), with 50 Gy in 25 daily fractions (2 Gy/fraction, 5 fractions weekly) for 5 weeks (week 1 - week 5).
  Arms: Neoadjuvant RT and ADT
Drug: Goserelin 3.6 MG — Gosereline 3.6mg sc injection at week 1, week 5, and week 9
  Other Names: ZOLADEX
Procedure: radical prostatectomy — Eligible patients will undergo robotic-assisted radical prostatectomy and pelvic lymph node dissection

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Androgens can stimulate the growth of prostate cancer cells. Hormone therapy can fight prostate cancer by androgen deprivation. It is not yet known if neoadjuvant radiation therapy is a more effective therapy for high-risk prostate cancer.

PURPOSE: Two-stage randomized trial to compare the effectiveness and safety of neoadjuvant radiotherapy and hormone therapy followed by radical prostatectomy in men with high-risk locally advanced prostate cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Success rate of salvage radiation therapy (SRT) measured as pathologic complete response (pCR) or pathologic near complete response (minimal residual disease, MRD) rate.

SECONDARY OBJECTIVES:

I. PSA decline rate after neoadjuvant treatment, rate of undetectable PSA after RP, rate of positive surgical margin, and rate of pathologic down-staging (≤ ypT2N0) II. Biochemical recurrence-free survival rate (from date of randomization). III. Metastasis free survival. IV. Prostate Cancer Death. V. Overall Survival

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive neoadjuvant hormone and radiation therapy, and then radical prostatectomy

ARM II: Participants receive neoadjuvant hormone therapy, and then radical prostatectomy.

After intervention, participants are followed up periodically for up to 20 years.

ELIGIBILITY:
Inclusion Criteria:

* Men with age from 20 to 75 years old
* Signed an informed consent form (ICF) indicating that the subject understands the purpose of and procedures required for the study and is willing to participate in the study; subjects must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Histologically confirmed adenocarcinoma of the prostate
* High-risk locally advanced disease defined by ≥1 of the following 3 criteria:

  * T3a-3b by DRE or MRI
  * Gleason score ≥ 8 (= Grade group 4)
  * PSA ≥20 ng/ml
* Willing to undergo prostatectomy as primary treatment
* ECOG Performance status 0 or 1

Exclusion Criteria:

* Pathological finding of small cell, ductal or neuroendocrine carcinoma
* Current or prior hormone therapy, radiotherapy, or chemotherapy
* Evidence of metastasis (M1) on images
* Other prior malignancy ≤5 years prior to enrollment
* Any of the following within 6 months prior to first dose of study drug: severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (eg, pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias or New York Heart Association Class II to IV heart disease; uncomplicated deep vein thrombosis is not considered exclusionary
* Human immunodeficiency virus-positive subjects with 1 or more of the following:

  1. Not receiving highly active antiretroviral therapy
  2. Had a change in antiretroviral therapy within 6 months of the start of screening
  3. Receiving antiretroviral therapy that may interfere with study drug (consult sponsor for review of medication prior to enrollment)
  4. CD4 count <350 at screening
  5. AIDS-defining opportunistic infection within 6 months of start of screening
* Active or symptomatic viral hepatitis or chronic liver disease; ascites or bleeding disorders secondary to hepatic dysfunction
* History of seizure or any condition that may predispose to seizure (including, but not limited to, prior stroke, transient ischemic attack, or loss of consciousness ≤1 year prior to randomization; brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect)
* Gastrointestinal conditions affecting absorption

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2041-07-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic outcome | From date of randomization to the date of radical prostatectomy, up to 100 weeks
  pathologic complete response (pCR) or pathologic near complete response (minimal residual disease, MRD) rate

SECONDARY OUTCOMES:
PSA decline percentage | From date of randomization to 10 years
  PSA decline is defined as nadir PSA value/baseline PSA value × 100
PSA complete response rate | From date of randomization to 10 years
  Complete response is defined as a drop in PSA on protocol treatment to less than 0.2 ng/ml.
PSA Recurrence | From date of randomization to 10 years
  Biochemical recurrence is defined as a rise in PSA to 0.2 ng/mL and a confirmatory value of 0.2 ng/mL or greater following radical prostatectomy
Distant Failure | From date of randomization to 10 years
  Distant failure rate is estimated by the cumulative incidence method, with failure defined as the first occurrence of distant failure.
Prostate Cancer Death | From date of randomization to 10 years
  Prostate cancer death rate us estimated by the cumulative incidence method, with failure defined as death due to prostate cancer or complications of trial.
Overall Survival | From date of randomization to 10 years
  Overall survival is estimated by the Kaplan-Meier method, with failure defined as death by any cause.
Progression-free Survival | From date of randomization to 10 years
  Progress-free survival is estimated by the Kaplan-Meier method, with failure defined as the first occurrence of PSA failure, local, regional or distant failure, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Yuan Huang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital Yunlin Branch, Douliu City/Huwei Township, Yunlin County
  - National Taiwan University Hospital, Tapiei

IPD SHARING:
Plan to Share IPD: No